CLINICAL TRIAL: NCT01399840
Title: Phase 1, Two-arm, Open-label Study Of Once Daily, Oral Bmn 673 In Patients With Advanced Hematological Malignancies
Brief Title: Study of BMN 673, a PARP Inhibitor, in Patients With Advanced Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP-002; 2010-023964-42 (EudraCT Number); C3441022 (Other: Alias Study Number)
Record Dates: First submitted 2011-07-13; First posted 2011-07-22 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — talazoparib

ARMS (2):
- Arm 1: BMN 673 (Experimental): Arm 1 will enroll patients with either AML or MDS
  Interventions: Drug: BMN 673
- Arm 2: BMN 673 (Experimental): Arm 2 will enroll patients with either CLL or MCL
  Interventions: Drug: BMN 673

INTERVENTIONS:
Drug: BMN 673 — Oral capsule with multiple dosage forms given once daily

SUMMARY:
This is a two-arm, open-label study to determine the maximum tolerated dose (MTD) and assess the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of BMN 673 in patients with Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS), Chronic Lymphocytic Leukemia (CLL) and Mantle Cell Lymphoma (MCL). Arm 1 will enroll patients with either AML or MDS; Arm 2 will enroll patients with either CLL or MCL.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
3. Arm 1 AML/MDS: Must have available tissue
4. Arm 2 CLL/MCL: Must have available tissue
5. Have adequate organ function as defined below:

   1. Serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 X upper limit of normal (ULN);
   2. Total serum bilirubin ≤ 1.5 X ULN;
6. Able to take oral medications
7. Recovered from acute toxicity of prior treatment
8. Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
9. If sexually active, must be willing to use an acceptable method of contraception during therapy and for 30 days after the last dose of BMN 673.
10. If female of childbearing potential, must have a negative serum pregnancy test at screening and be willing to have additional pregnancy tests during the study.
11. Willing and able to comply with all study procedures.

Exclusion Criteria:

1. Acute promyelocytic leukemia, APL [AML with t(15;17)(q22;q12), PML-RARA and variants].
2. Disease-specific exclusion criteria:

   a. AML: i. Marrow cellularity < 25% ii. Circulating blasts > 50,000/mm3 b. MCL and CLL: i. Platelet count < 50,000/mm3 ii. Neutrophil count < 1000/mm3
3. Autologous bone marrow transplant < 6 months before Cycle 1 Day 1
4. Prior allogeneic bone marrow transplant < 6 months before Cycle 1 Day 1 and/or with the presence of graft versus host disease (GVHD)
5. Prior treatment:

   1. AML: anti-leukemia treatment within 14 days before Cycle 1 Day 1; hydroxyurea treatment within 7 days before Cycle 1 Day 1.
   2. CLL, MCL or MDS: anti-lymphoma/leukemia treatment within 28 days before Cycle 1 Day 1;
6. CLL/MCL patients who have received transfusion, hematopoietic growth factors within 7 days before Cycle 1 Day 1.
7. Symptomatic central nervous system (CNS) involvement.
8. Known to have human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or hepatitis B virus (HBV).
9. Major surgery within 28 days before Cycle 1, Day 1.
10. Active peptic ulcer disease.
11. Active gastrointestinal tract disease with malabsorption syndrome.
12. Requirement for IV alimentation.
13. Prior surgical procedures affecting absorption.
14. Uncontrolled inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
15. Myocardial infarction within 6 months before Cycle 1 Day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication.
16. Breastfeeding at screening or planning to become pregnant (self or partner) at any time during study participation.
17. Use of any investigational product or investigational medical device within 28 days before Cycle 1, Day 1.
18. Concurrent disease or condition that would interfere with study participation or safety, such as:

    1. CLL/MCL patients with active, clinically significant infection requiring the use of parenteral anti-microbial agents, or grade > 2 infection by NCI CTCAE (v4.03) within 14 days before Cycle 1, Day 1(AML/MDS patients with controlled infection are eligible for the study with no specific time requirement prior to Cycle 1, Day 1);
    2. Clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders;
    3. Non-healing wound, ulcer, or bone fracture.
19. Patients who have received prior treatment with a PARP inhibitor are not eligible for Part 2 of the study (expansion), but are eligible for Part 1 (dose escalation) of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-05-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is to determine the MTD of daily oral BMN 673 in patients with AML and MDS (Arm 1) and patients with CLL and MCL (Arm 2). | Assessed after each visit until completion (Estimated duration is 12-18 months)

SECONDARY OUTCOMES:
Number of participants with adverse events | Assessed after each visit until completion of the study (Estimated duration is 24-30 months)
Determine the pharmacokinetic (PK) profile of BMN 673 | Assessed at each visit in cycle 1 - 5 (Estimated duration is 24 months)
  Sample collection times vary per visit. PK parameters that will be evaluated include: maximum concentration (Cmax), minimum concentration (Cmin), time to maximum plasma concentration (Tmax), area under the curve from 0 to last quantifiable sampling point postdose (AUC0-inf), area under the curve extrapolated to infinity (AUC0-last), half life (t1/2), systemic clearance (CL/f) and volume of ditribution (VZ/f)
Determine the Recommended Phase 2 Dose (RP2D) of oral daily BMN 673 | Assessed after each visit until completion of the study (Estimated duration is 24-30 months)
Assess preliminary efficacy of BMN 673 by evaluating per response publications | Assessed approximately every 4-12 weeks (Estimated duration is 24-30 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (3):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- United Kingdom (4):
  - University College London, London
  - King's College Hospital, London
  - The Christie NHS Foundation, Manchester
  - University of Newcastle Upon Tyne, NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Gopal AK, Popat R, Mattison RJ, Menne T, Bloor A, Gaymes T, Khwaja A, Juckett M, Chen Y, Cotter MJ, Mufti GJ. A Phase I trial of talazoparib in patients with advanced hematologic malignancies. Int J Hematol Oncol. 2021 Oct 22;10(3):IJH35. doi: 10.2217/ijh-2021-0004. eCollection 2021 Sep. PMID 34840720